CLINICAL TRIAL: NCT00501826
Title: Phase II Study of Hyper-CVAD Plus Nelarabine in Previously Untreated T-ALL and Lymphoblastic Lymphoma
Brief Title: Combination Chemotherapy and Nelarabine in Treating Patients With T-cell Acute Lymphoblastic Leukemia or Lymphoblastic Lymphoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Purpose: Treatment
Other Study IDs: 2006-0328; NCI-2012-01518 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2006-0328 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2007-07-12; First posted 2007-07-16 (Estimated); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: T Acute Lymphoblastic Leukemia; T Lymphoblastic Lymphoma
MeSH Terms: conditions — Precursor T-Cell Lymphoblastic Leukemia-Lymphoma | interventions — Cyclophosphamide; Cytarabine; Dexamethasone; Calcium Dobesilate; auricularum; dexamethasone acetate; dexamethasone 21-phosphate; Doxorubicin; Mercaptopurine; azathiopurine; Methotrexate; merphos; nelarabine; pegaspargase; Prednisone; deltacortene; prednylidene; venetoclax; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (nelarabine and combination chemotherapy) (Experimental): See Detailed Description
  Interventions: Drug: Cyclophosphamide; Drug: Cytarabine; Drug: Dexamethasone; Drug: Doxorubicin Hydrochloride; Drug: Mercaptopurine; Drug: Methotrexate; Drug: Nelarabine; Drug: Pegaspargase; Drug: Prednisone; Drug: Venetoclax; Drug: Vincristine Sulfate

INTERVENTIONS:
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719
Drug: Cytarabine — Given IV
  Other Names: .beta.-Cytosine arabinoside; 1-.beta.-D-Arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-.beta.-D-Arabinofuranosylcytosine; 1-Beta-D-arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-Beta-D-arabinofuranosylcytosine; 1.beta.-D-Arabinofuranosylcytosine; 2(1H)-Pyrimidinone, 4-Amino-1-beta-D-arabinofuranosyl-; 2(1H)-Pyrimidinone, 4-amino-1.beta.-D-arabinofuranosyl-; Alexan; Ara-C; ARA-cell; Arabine; Arabinofuranosylcytosine; Arabinosylcytosine; Aracytidine; Aracytin; Aracytine; Beta-cytosine Arabinoside; CHX-3311; Cytarabinum; Cytarbel; Cytosar; Cytosine Arabinoside; Cytosine-.beta.-arabinoside; Cytosine-beta-arabinoside; Erpalfa; Starasid; Tarabine PFS; U 19920; U-19920; Udicil; WR-28453
Drug: Dexamethasone — Given IV or PO
  Other Names: Aacidexam; Adexone; Aknichthol Dexa; Alba-Dex; Alin; Alin Depot; Alin Oftalmico; Amplidermis; Anemul mono; Auricularum; Auxiloson; Baycadron; Baycuten; Baycuten N; Cortidexason; Cortisumman; Decacort; Decadrol; Decadron; Decadron DP; Decalix; Decameth; Decasone R.p.; Dectancyl; Dekacort; Deltafluorene; Deronil; Desamethasone; Desameton; Dexa-Mamallet; Dexa-Rhinosan; Dexa-Scheroson; Dexa-sine; Dexacortal; Dexacortin; Dexafarma; Dexafluorene; Dexalocal; Dexamecortin; Dexameth; Dexamethasone Intensol; Dexamethasonum; Dexamonozon; Dexapos; Dexinoral; Dexone; Dinormon; Fluorodelta; Fortecortin; Gammacorten; Hexadecadrol; Hexadrol; Lokalison-F; Loverine; Methylfluorprednisolone; Millicorten; Mymethasone; Orgadrone; Spersadex; TaperDex; Visumetazone; ZoDex
Drug: Doxorubicin Hydrochloride — Given IV
  Other Names: 5,12-Naphthacenedione, 10-[(3-amino-2,3,6-trideoxy-alpha-L-lyxo-hexopyranosyl)oxy]-7,8, 9,10-tetrahydro-6,8,11-trihydroxy-8-(hydroxyacetyl)-1-methoxy-, hydrochloride, (8S-cis)- (9CI); ADM; Adriacin; Adriamycin; Adriamycin Hydrochloride; Adriamycin PFS; Adriamycin RDF; ADRIAMYCIN, HYDROCHLORIDE; Adriamycine; Adriblastina; Adriblastine; Adrimedac; Chloridrato de Doxorrubicina; DOX; DOXO-CELL; Doxolem; Doxorubicin HCl; Doxorubicin.HCl; Doxorubin; Farmiblastina; FI 106; FI-106; hydroxydaunorubicin; Rubex
Drug: Mercaptopurine — Given PO
  Other Names: 3H-Purine-6-thiol; 6 MP; 6 Thiohypoxanthine; 6 Thiopurine; 6-Mercaptopurine; 6-Mercaptopurine Monohydrate; 6-MP; 6-Purinethiol; 6-Thiopurine; 6-Thioxopurine; 6H-Purine-6-thione, 1,7-dihydro- (9CI); 7-Mercapto-1,3,4,6-tetrazaindene; Alti-Mercaptopurine; Azathiopurine; BW 57-323H; Flocofil; Ismipur; Leukerin; Leupurin; Mercaleukim; Mercaleukin; Mercaptina; Mercaptopurinum; Mercapurin; Mern; NCI-C04886; Puri-Nethol; Purimethol; Purine, 6-mercapto-; Purine-6-thiol (8CI); Purine-6-thiol, monohydrate; Purinethiol; Purinethol; U-4748; WR-2785
Drug: Methotrexate — Given IV and PO
  Other Names: Abitrexate; Alpha-Methopterin; Amethopterin; Brimexate; CL 14377; CL-14377; Emtexate; Emthexat; Emthexate; Farmitrexat; Fauldexato; Folex; Folex PFS; Lantarel; Ledertrexate; Lumexon; Maxtrex; Medsatrexate; Metex; Methoblastin; Methotrexate LPF; Methotrexate Methylaminopterin; Methotrexatum; Metotrexato; Metrotex; Mexate; Mexate-AQ; MTX; Novatrex; Rheumatrex; Texate; Tremetex; Trexeron; Trixilem; WR-19039
Drug: Nelarabine — Given IV
  Other Names: 2-Amino-6-methoxypurine arabinoside; 506U78; Arranon; Compound 506U78; GW506U78
Drug: Pegaspargase — Given IV
  Other Names: L-Asparaginase with Polyethylene Glycol; Oncaspar; Oncaspar-IV; PEG-Asparaginase; PEG-L-Asparaginase; PEG-L-Asparaginase (Enzon - Kyowa Hakko); PEGLA; Polyethylene Glycol L-Asparaginase; Polyethylene Glycol-L-Asparaginase
Drug: Prednisone — Given PO
  Other Names: .delta.1-Cortisone; 1, 2-Dehydrocortisone; Adasone; Cortancyl; Dacortin; DeCortin; Decortisyl; Decorton; Delta 1-Cortisone; Delta-Dome; Deltacortene; Deltacortisone; Deltadehydrocortisone; Deltasone; Deltison; Deltra; Econosone; Lisacort; Meprosona-F; Metacortandracin; Meticorten; Ofisolona; Orasone; Panafcort; Panasol-S; Paracort; Perrigo Prednisone; PRED; Predicor; Predicorten; Prednicen-M; Prednicort; Prednidib; Prednilonga; Predniment; Prednisone Intensol; Prednisonum; Prednitone; Promifen; Rayos; Servisone; SK-Prednisone
Drug: Venetoclax — Given PO
  Other Names: ABT-0199; ABT-199; ABT199; GDC-0199; RG7601; Venclexta; Venclyxto
Drug: Vincristine Sulfate — Given IV
  Other Names: Kyocristine; Leurocristine sulfate; Leurocristine, sulfate; Oncovin; Vincasar; Vincosid; Vincrex; Vincristine, sulfate

SUMMARY:
This phase II trial studies the side effects and how well combination chemotherapy and nelarabine work in treating patients with T-cell acute lymphoblastic leukemia or lymphoblastic lymphoma. Drugs used in chemotherapy, such as cyclophosphamide, vincristine, doxorubicin, dexamethasone, methotrexate, cytarabine, mercaptopurine, prednisone, pegaspargase, nelarabine, and venetoclax work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the complete remission (CR) rate and progression-free survival following treatment with hyperfractionated cyclophosphamide, vincristine sulfate, doxorubicin hydrochloride, and dexamethasone (hyper-CVAD) in combination with nelarabine in previously untreated patients with T-cell acute lymphoblastic leukemia (ALL) and T-cell lymphoblastic lymphoma.

II. To determine the safety and overall survival of previously untreated patients with T-cell ALL and T-cell lymphoblastic lymphoma.

III. To determine the safety and efficacy of adding pegaspargase to the regimen.

IV. To determine the safety and efficacy of adding venetoclax to the regimen.

OUTLINE:

COURSES 1, 3, 5, and 7 (hyper-CVAD): Patients receive cyclophosphamide intravenously (IV) over 3 hours twice daily (BID) on day 1-3, doxorubicin IV over 24 hours on day 4, vincristine IV over 15-30 minutes on days 4 and 11, and dexamethasone IV or orally (PO) once daily (QD) on days 1-4 and 11-14.

COURSES 2, 4, 6, and 8 (methotrexate/cytarabine): Patients receive methotrexate IV over 24 hours on day 1 and cytarabine IV over 2 hours BID on days 2 and 3.

Patients also receive venetoclax PO QD on days 1-14 of each course. Courses of hyper-CVAD and methotrexate/cytarabine repeat every 21 days in the absence of disease progression or unacceptable toxicity.

Patients also receive nelarabine IV over 2 hours once daily (QD) for 5 days and pegaspargase IV over 2 hours on day 5 after completion of course 4 and after the completion of course 5 in the absence of disease progression or unacceptable toxicity.

MAINTENANCE COURSES 1-5, 8-17, and 20-30 (mercaptopurine, vincristine, methotrexate, and prednisone [POMP]): Patients receive mercaptopurine PO thrice daily (TID), methotrexate PO once weekly, vincristine sulfate IV on day 1, prednisone PO QD on days 1-5, and venetoclax PO QD on days 1-7. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

INTENSIFICATION COURSES 6 and 7: Patients receive nelarabine IV QD over 2 hours on days 1-5 and pegaspargase IV over 2 hours on day 5. Patients also receive venetoclax PO QD on days 1-14. Courses repeat every 21-35 days in the absence of disease progression or unacceptable toxicity.

INTENSIFICATION COURSES 18 and 19: Patients receive methotrexate IV over 2 hours on day 1, pegaspargase IV over 2 hours on day 2, and venetoclax PO QD on days 1-14 in the absence of disease progression or unacceptable toxicity.

POMP maintenance therapy continues for 30 months in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3-6 months.

ELIGIBILITY:
Inclusion Criteria:

* Previously untreated T cell ALL including T cell lymphoblastic lymphoma; failure to one induction course of chemotherapy are eligible; patients in CR after =< 2 courses are also eligible
* Eastern Cooperative Oncology Group (ECOG) performance status less than or equal to 3
* Serum bilirubin less than or equal to 2.0 mg/dL unless considered due to involvement by tumor when an upper limit of 5.0 mg/dL is acceptable
* Serum glutamic oxaloacetic transaminase (SGOT) or serum glutamate pyruvate transaminase (SGPT) less than or equal to 4 x upper limit of normal (ULN)
* Serum creatinine less than or equal to 2.0 mg/dL unless considered due to involvement by tumor when an upper limit of 2.5 mg/dL is acceptable

Exclusion Criteria:

* Pregnant or nursing women

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2007-07-11 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Complete remission rate | 3 years
  The sample size will provide an estimate of relapse rate at 3 years with a 95% confidence interval of width +/- 10%.
Duration of remission | Up to 9 years
  Duration of remission will be evaluated.
Progression-free survival | 3 years
  Progression-free survival will be estimated.
Overall survival | 3 years
  Overall survival will be estimated.

CONTACTS AND LOCATIONS:
Overall Officials: Farhad Ravandi-Kashani, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org